CLINICAL TRIAL: NCT02887937
Title: Qualitative and Quantitative Analysis of Cystic Breast Masses by Contrast Enhanced Ultrasound: Is Biopsy Necessary?
Brief Title: Cystic Breast Masses by Contrast Enhanced Ultrasound (CEUS)
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Wright Foundation (Unknown)
Responsible Party: Principal Investigator, Sandy Lee, Assistant Professor, University of Southern California
Other Study IDs: HS-16-00483
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — perflutren

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Breast Mass 4a-cystic: Contrast Enhanced UltraSound (CEUS) exams will be performed on a ultrasound machine for the 4a-cystic breast masses recommended for biopsy. An intravenous line (IV) line will be inserted into the vein in the arm for the administration of the contrast agent, Definity (10 µL/kg) The patient will be asked to lie on a table for the 4DCT and unenhanced CT procedure and the images will be recorded. For the contrast enhanced ultrasound, the contrast agent will be injected into the IV line. The CEUS will be performed and the images will be recorded. The contrast agent may be administered two to three more times as needed. Scanning will then be repeated with 30 and 90 seconds delay after the IV contrast administration.
  Interventions: Drug: Definity
- Breast Mass 4a- non cystic: Contrast Enhanced UltraSound (CEUS) exams will be performed on a ultrasound machine for the 4a-non cystic breast masses recommended for biopsy. An intravenous line (IV) line will be inserted into the vein in the arm for the administration of the contrast agent, Definity (10 µL/kg) The patient will be asked to lie on a table for the 4DCT and unenhanced CT procedure and the images will be recorded. For the contrast enhanced ultrasound, the contrast agent will be injected into the IV line. The CEUS will be performed and the images will be recorded. The contrast agent may be administered two to three more times as needed. Scanning will then be repeated with 30 and 90 seconds delay after the IV contrast administration..
  Interventions: Drug: Definity
- Breast Mass 4b: Contrast Enhanced UltraSound (CEUS) exams will be performed on a ultrasound machine for the 4b breast masses recommended for biopsy. An intravenous line (IV) line will be inserted into the vein in the arm for the administration of the contrast agent, Definity (10 µL/kg) The patient will be asked to lie on a table for the 4DCT and unenhanced CT procedure and the images will be recorded. For the contrast enhanced ultrasound, the contrast agent will be injected into the IV line. The CEUS will be performed and the images will be recorded. The contrast agent may be administered two to three more times as needed. Scanning will then be repeated with 30 and 90 seconds delay after the IV contrast administration.
  Interventions: Drug: Definity
- Breast Mass 4c: Contrast Enhanced UltraSound (CEUS) exams will be performed on a ultrasound machine for the 4c breast masses recommended for biopsy. An intravenous line (IV) line will be inserted into the vein in the arm for the administration of the contrast agent, Definity (10 µL/kg) The patient will be asked to lie on a table for the 4DCT and unenhanced CT procedure and the images will be recorded. For the contrast enhanced ultrasound, the contrast agent will be injected into the IV line. The CEUS will be performed and the images will be recorded. The contrast agent may be administered two to three more times as needed. Scanning will then be repeated with 30 and 90 seconds delay after the IV contrast administration.
  Interventions: Drug: Definity

INTERVENTIONS:
Drug: Definity — The contrast agent, Definity, 10 µL/kg, will be administered through an intravenous catheter placed in an antecubital vein. Definity is an FDA approved contrast agent for cardiac studies and will be an off-label use in this study. The agent will be injected as a single intravenous bolus followed by a 10 mL saline flush (0.9% NaCl). Images will be recorded with clip function for 90 seconds following the administration of contrast while the probe is stabilized and minimal pressure applied. During this time, qualitative evaluation of tumor enhancement will be observed, and the presence of contrast uptake within the tumor will be categorized.
  Other Names: Perflutren

SUMMARY:
The overarching goal of the proposed research is to evaluate whether qualitative and quantitative parameters in real time contrast enhanced ultrasound (CEUS) can aid in assessing suspicious indeterminate cystic appearing breast masses and ultimately determine whether or not an ultrasound guided biopsy is necessary. The underlying hypothesis is that breast masses (given BIRADS 4) that lack enhancement on CEUS will have a benign histology obtained by ultrasound guided core biopsy and/or surgery. Then, in the future, these non-enhancing cystic lesions can be followed and do not need biopsy intervention.

DETAILED DESCRIPTION:
Breast cancer is the most frequently diagnosed cancer in women. To diagnose these cancers, more than 1.6 million breast biopsies are performed each year in the United States, of which more than 60% have benign pathology. A large percentage of the benign biopsies show fibrocystic changes of the breast on histology. These biopsies can be avoided with better diagnostic tools identifying fibrocystic change. The Investigators propose that contrast enhanced ultrasound (CEUS) can aid in classifying and predicting if a cystic appearing breast mass is benign or malignant, and can be a supplemental imaging tool to mammography and conventional gray-scale ultrasound (US).

In standard clinical practice, if a breast mass appears to be cystic on gray-scale US but has some suspicious features which make it difficult to tell if the mass is truly cystic or solid, the decision making for follow-up versus biopsy is difficult. This leads to unnecessary biopsies (false positives) since many of these masses are a sequel of benign fibrosis and fibrocystic changes of the breast. CEUS may help classify these masses as cystic or solid. The central premise is based on the microbubble contrast agent used in CEUS, since it stays within the blood pool and will only show enhancement if a mass has solid components and has vascular flow.

The Investigators hypothesize that indeterminate cystic breast masses will not enhance on CEUS and will correlate with benign pathology. Quantitative CEUS parameters will also help classify these lesions. If this is the case, then in the future, the non-enhancing cystic breast masses will not need to be biopsied. This will decrease patient anxiety, unnecessary interventions, and save resources.

The investigators will investigate qualitative and quantitative parameters on CEUS in evaluating indeterminate cystic breast masses given BIRADS 4 and correlate these with histopathology obtained by biopsy and/or surgery. This data will help them to develop protocols to better distinguish between benign and malignant cystic appearing breast masses.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* recommended for an ultrasound guided biopsy due to breast mass detection

Exclusion Criteria:

* < 18 years of age
* prior history of breast cancer
* prior history of biopsy for that specific lesion
* any condition that would be a contraindication to the microbubble contrast agent used in CEUS such as pulmonary hypertension, 3cardiac shunts, and allergy to perflutren.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will be performed as a prospective study at LAC+USC in the mammography department. Our project will enroll approximately 135 women > 18 years of age with breast masses evaluated by conventional US given BIRADS 4 and recommended for ultrasound guided biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2018-04-29 (Actual)

PRIMARY OUTCOMES:
lesions of malignant vs. benign biopsy histology | 0-2 months
  The proportion of breast masses with presence of contrast uptake on CEUS will be calculated for lesions of malignant vs. benign biopsy histology, grouped by BIRADS categories

SECONDARY OUTCOMES:
classification rule with the CEUS parameters | 11-12 months
  We will build a classification rule with the CEUS parameters and then assess whether this rule can classify benign or malignant BIRADS 4a cystic lesions correctly.

CONTACTS AND LOCATIONS:
Overall Officials: Sandy C Lee, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Department of Radiology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided